CLINICAL TRIAL: NCT01217892
Title: A 16-week, Multicentre, Randomised, Double-Blind, Placebo-Controlled Phase III Study to Evaluate the Safety and Efficacy of Dapagliflozin 2.5 mg BID, 5 mg BID and 10 mg QD Versus Placebo in Patients With Type 2 Diabetes Who Are Inadequately Controlled on Metformin-IR Monotherapy
Brief Title: Evaluation of Dapagliflozin Taken Twice-daily
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1691C00003
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; metformin treated; inadequate control; metformin treatment alone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Dapagliflozin 2.5 mg twice-daily plus open-label metformin
  Interventions: Drug: dapagliflozin; Drug: metformin
- 2 (Experimental): Dapagliflozin 5.0 mg twice-daily plus open-label metformin
  Interventions: Drug: dapagliflozin; Drug: metformin
- 3 (Experimental): Dapagliflozin 10 mg once-daily plus open-label metformin
  Interventions: Drug: dapagliflozin; Drug: metformin
- 4 (Placebo Comparator): Placebo plus open-label metformin
  Interventions: Drug: metformin; Drug: placebo

INTERVENTIONS:
Drug: dapagliflozin — 2.5 mg tablet, taken orally, twice daily
  Arms: 1
Drug: dapagliflozin — 5 mg tablet taken orally, twice daily
  Arms: 2
Drug: dapagliflozin — 10 mg tablet taken orally, once daily
  Arms: 3
Drug: metformin — >/= 1500 mg total daily dose, tablets taken orally, twice daily
Drug: placebo — placebo
  Arms: 4

SUMMARY:
This study is being carried out to see if dapagliflozin - administered in a daily dose of 2.5 mg given twice a day or 5 mg twice a day or 10mg once daily - in addition to metformin, is beneficial in diabetes treatment, and if so, how it compares to treatment with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Diagnosis of T2DM
* Current antihyperglycaemic treatment with metformin immediate release formulation monotherapy >/= 1500 mg/day at a stable dose for at least 10 weeks prior to enrolment. Other treatment with OADs within the 10 weeks prior to enrolment is not permitted.
* HbA1c ≥ 6.7% and ≤10.5%, based on central laboratory values from Screening Visit, and Enrolment Visit 1.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus, known diagnosis of Maturity Onset Diabetes of the Young (MODY) or secondary causes of diabetes mellitus
* History of diabetic ketoacidosis
* Symptoms of poorly controlled diabetes including, but not limited to, marked polyuria, polydipsia, and/or greater than 10% weight loss during the 3 months prior to enrolment
* FPG >270 mg/dL (>15.0 mmol/L)
* BMI >45 kg/m2

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Parikh, Study Director — AstraZeneca
Locations (55):
- Germany (11):
  - Research Site, Aßlar
  - Research Site, Berlin
  - Research Site, Biberach A.d. Riss
  - Research Site, Bosenheim
  - Research Site, Dippoldiswalde
  - Research Site, Falkensee
  - Research Site, Meissen
  - Research Site, München
  - Research Site, Neuwied
  - Research Site, Pirna
  - Research Site, Wahlstedt
- Hungary (10):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Csongrád
  - Research Site, Debrecen
  - Research Site, Gyöngyös
  - Research Site, Kecskemét
  - Research Site, Makó
  - Research Site, Nyíregyháza
  - Research Site, Tát
  - Research Site, Zalaegerszeg
- Romania (5):
  - Research Site, Brasov, Brașov County
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Sibiu
  - Research Site, Suceava
- Slovakia (11):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Námestovo
  - Research Site, Piešťany
  - Research Site, Prievidza
  - Research Site, Rimavská Sobota
  - Research Site, Ružomberok
  - Research Site, Žilina
- South Africa (6):
  - Research Site, Verulam, KwaZulu-Natal
  - Research Site, Cape Town, South Africa
  - Research Site, Durban, South Africa
  - Research Site, eMkhomazi, South Africa
  - Research Site, Johannesburg, South Africa
  - Research Site, Durban
- Switzerland (7):
  - Research Site, Chur, Kanton Graubünden
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Kreuzlingen
  - Research Site, Lugano
  - Research Site, Rorschach
- Ukraine (5):
  - Research Site, Vynnitsa, Ukraine
  - Research Site, Zaporizhzhya, Ukraine
  - Research Site, Dnipropetrov'sk
  - Research Site, Kiev
  - Research Site, Vinnytsia

REFERENCES:
- [Background] Schumm-Draeger PM, Burgess L, Koranyi L, Hruba V, Hamer-Maansson JE, de Bruin TW. Twice-daily dapagliflozin co-administered with metformin in type 2 diabetes: a 16-week randomized, placebo-controlled clinical trial. Diabetes Obes Metab. 2015 Jan;17(1):42-51. doi: 10.1111/dom.12387. Epub 2014 Oct 16. PMID 25200570
- See also: CSR-D1691C00003.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=296&filename=CSR-D1691C00003.pdf
- See also: D1691C00003_Clinical_Study_Protocol_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=296&filename=D1691C00003_Clinical_Study_Protocol_Redacted_10Jun2014.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 5 November 2010. Last participant last visit for the 16-week period: 25 August 2011. 520 participants were enrolled, and 400 were randomized in 53 study centers in Europe and South Africa. Subjects with T2DM who showed inadequate glycemic control on metformin therapy alone.
Pre-assignment Details: During a placebo lead-in period, participants were counselled on dietary and life-style modifications. Subjects eligible for the study were stratified according to their baseline HbA1c.
Groups:
- Dapagliflozin 2.5mg BID Plus Metformin: Dapagliflozin 2.5mg, oral, twice daily plus Metformin, oral, twice daily, >=1500mg total daily dose
- Dapagliflozin 5mg BID Plus Metformin: Dapagliflozin 5mg, oral, twice daily plus Metformin, oral, twice daily, >=1500mg total daily dose
- Dapagliflozin 10mg OD Plus Metformin: Dapagliflozin 10mg, oral, once daily plus Metformin, oral, twice daily, >=1500mg total daily dose
- Placebo Plus Metformin: Placebo plus Metformin, oral, twice daily, >=1500mg total daily dose
Period: Overall Study
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin
Started | 100 | 100 | 99 | 101
Completed | 93 | 94 | 90 | 93
Not Completed | 7 | 6 | 9 | 8
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0
Not completed — Lab value | 1 | 0 | 1 | 0
Not completed — Subject no longer meets study criteria | 5 | 2 | 4 | 8
Not completed — Incorrect enrollment | 0 | 1 | 1 | 0
Not completed — Poor/Non-Compliance | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin | Total
Number analyzed (Participants) | 100 | 99 | 99 | 101 | 399
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (9.01) | 55.3 (9.34) | 58.5 (9.78) | 58.5 (9.40) | 57.7 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 53 | 50 | 54 | 220
  Male | 37 | 46 | 49 | 47 | 179
HbA1c [Mean (Standard Deviation); unit: Percent [%]] | 7.77 (0.747) | 7.78 (0.762) | 7.71 (0.709) | 7.94 (0.848) | 7.80 (0.770)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 153.3 (33.27) | 155.3 (31.92) | 155.3 (36.26) | 157.8 (35.93) | 155.4 (34.30)
Body weight [Mean (Standard Deviation); unit: kg] | 92.49 (18.632) | 93.62 (16.641) | 90.58 (15.929) | 88.82 (15.327) | 91.37 (16.716)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To compare the change from baseline in HbA1c achieved with each of the 2 BID doses of dapagliflozin (2.5 mg BID and 5 mg BID) co-administered with metformin versus placebo co-administered with metformin after 16 weeks of double-blind treatment.
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and Week 16 (LOCF) values
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin
Number analyzed (Participants) | 99 | 97 | 98 | 100
Percent | -0.52 (0.0594) [-0.63 to -0.40] | -0.65 (0.0600) [-0.77 to -0.53] | -0.59 (0.0598) [-0.70 to -0.47] | -0.30 (0.0593) [-0.42 to -0.18]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg BID Plus Metformin vs Placebo Plus Metformin; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0 (with alpha = 0.05 using Hochberg's method to control the overall Type I error across hypotheses in the two Dapagliflozin BID groups, two-sided); Test type: Superiority or Other; p = 0.0106, ANCOVA — significant at alpha=0.05 (2-sided) applying Hochberg's method across the two Dapagliflozin BID groups; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.38 to -0.05], Standard Error of Mean 0.0840
Statistical Analysis 2: Comparison: Dapagliflozin 5mg BID Plus Metformin vs Placebo Plus Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.05 (2-sided) applying Hochberg's method across the two Dapagliflozin BID groups; with treatment group as effect (all treatment groups included) and baseline value as covariate; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.52 to -0.18], Standard Error of Mean 0.0843

2. Secondary Outcome: Adjusted Percent Change in Body Weight
Description: To compare the percent change from baseline in body weight achieved with each of the 2 BID doses of dapagliflozin (2.5 mg BID, and 5 mg BID) co-administered with metformin versus placebo co-administered with metformin after 16 weeks of double-blind treatment.
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and Week 16 (LOCF) values
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin
Number analyzed (Participants) | 100 | 99 | 99 | 101
Percent | -2.84 (0.3099) | -3.20 (0.3125) | -2.76 (0.3086) | -1.04 (0.3105)
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg BID Plus Metformin vs Placebo Plus Metformin; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0 (with alpha = 0.05, two-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.05 (2-sided). Key secondary endpoints are tested following a hierarchical closed testing procedure within treatment group for treatment groups tested significantly different from placebo for the primary endpoint; with treatment group (all treatment groups included) and stratum (HbA1c <7.0% vs >=7.0% at randomization) as effect and baseline value as covariate; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-2.53 to -1.10], Standard Error of Mean 0.3630
Statistical Analysis 2: Comparison: Dapagliflozin 5mg BID Plus Metformin vs Placebo Plus Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-2.89 to -1.46], Standard Error of Mean 0.3636

3. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose (FPG) From Baseline to Week 1
Description: To compare the change from baseline in fasting plasma glucose (FPG) achieved with each of the 2 BID doses of dapagliflozin (2.5 mg BID and 5 mg BID) co-administered with metformin versus placebo co-administered with metformin after 1 week of double-blind treatment.
Time Frame: Baseline to Week 1
Population: Full Analysis Set, participants with non-missing baseline and Week 1 values
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin
Number analyzed (Participants) | 99 | 99 | 98 | 101
mg/dL | -13.7 (2.657) | -14.7 (2.672) | -15.5 (2.634) | 2.0 (2.584)
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg BID Plus Metformin vs Placebo Plus Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -15.7, 95% CI 2-sided [-21.7 to -9.7], Standard Error of Mean 3.040
Statistical Analysis 2: Comparison: Dapagliflozin 5mg BID Plus Metformin vs Placebo Plus Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-22.7 to -10.7], Standard Error of Mean 3.039

4. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose (FPG) From Baseline to Week 16
Description: To compare the change from baseline in fasting plasma glucose (FPG) achieved with each of the 2 BID doses of dapagliflozin (2.5 mg BID and 5 mg BID) co-administered with metformin versus placebo co-administered with metformin after 16 weeks of double-blind treatment.
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and Week 16 (LOCF) values
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin
Number analyzed (Participants) | 100 | 99 | 98 | 101
mg/dL | -20.8 (2.738) | -25.6 (2.759) | -20.4 (2.720) | -10.4 (2.669)
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg BID Plus Metformin vs Placebo Plus Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0010, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-16.5 to -4.2], Standard Error of Mean 3.132
Statistical Analysis 2: Comparison: Dapagliflozin 5mg BID Plus Metformin vs Placebo Plus Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -15.3, 95% CI 2-sided [-21.4 to -9.1], Standard Error of Mean 3.139

5. Secondary Outcome: Proportion of Participants With HbA1c<7.0% at Week 16, in Participants Who Had HbA1c ≥7.0% at Baseline.
Description: To compare the adjusted proportions controlling for baseline HbA1c [acc. to Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu] of participants with HbA1c <7.0% achieved with each of the 2 BID doses of dapagliflozin (2.5 mg BID and 5 mg BID) co-administered with metformin versus placebo co-administered with metformin after 16 weeks of double-blind treatment, in patients who had HbA1c ≥7.0% at baseline.
Time Frame: Baseline to Week 16
Population: Full Analysis Set, participants with non-missing baseline and Week 16 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin
Number analyzed (Participants) | 89 | 90 | 81 | 87
Percentage of participants | 33.6 [24.6 to 42.5] | 38.2 [29.1 to 47.3] | 28.1 [19.0 to 37.1] | 21.4 [13.2 to 29.6]
Statistical Analysis 1: Comparison: Dapagliflozin 2.5mg BID Plus Metformin vs Placebo Plus Metformin; H0: proportion(treat) minus proportion(placebo) = 0 versus the alternative HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p = 0.0455, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = 12.2, 95% CI 2-sided [0.2 to 24.1], Standard Error of Mean 6.097
Statistical Analysis 2: Comparison: Dapagliflozin 5mg BID Plus Metformin vs Placebo Plus Metformin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0062, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = 16.8, 95% CI 2-sided [4.8 to 28.9], Standard Error of Mean 6.153

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 16 weeks double-blind treatment period plus 4 days / 30 days or up to follow-up visit if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Dapagliflozin 2.5mg BID Plus Metformin | Dapagliflozin 5mg BID Plus Metformin | Dapagliflozin 10mg OD Plus Metformin | Placebo Plus Metformin
Serious Adverse Events (participants affected / at risk) | 4/100 | 1/100 | 2/99 | 0/101
Other Adverse Events (participants affected / at risk) | 8/100 | 0/100 | 6/99 | 9/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 2.5mg BID Plus Metformin (N=100) | Dapagliflozin 5mg BID Plus Metformin (N=100) | Dapagliflozin 10mg OD Plus Metformin (N=99) | Placebo Plus Metformin (N=101)
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 | 0 | 0 | 0
ENDOMETRITIS (Infections and infestations) | 1 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 2.5mg BID Plus Metformin (N=100) | Dapagliflozin 5mg BID Plus Metformin (N=100) | Dapagliflozin 10mg OD Plus Metformin (N=99) | Placebo Plus Metformin (N=101)
INFLUENZA (Infections and infestations) | 5 | 0 | 2 | 3
HYPERTENSION (Vascular disorders) | 3 | 0 | 4 | 6

LIMITATIONS AND CAVEATS:
For participants who did not complete 16 weeks LOCF (last observation carried forward) was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.